CLINICAL TRIAL: NCT00495404
Title: Health Outcomes From Opioid Therapy for Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 98-149
Record Dates: First submitted 2007-06-29; First posted 2007-07-03 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-06

CONDITIONS: Chronic Pain; Behavior, Addictive
Keywords: chronic non-malignant pain; opiates; prescriptions; addiction
MeSH Terms: conditions — Chronic Pain; Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Other)
  Interventions: Behavioral: Physician Treatment Guidelines
- Arm 2 (Other)
  Interventions: Behavioral: Physician Treatment Guidelines

INTERVENTIONS:
Behavioral: Physician Treatment Guidelines

SUMMARY:
Although the use of opioid medications has gained increasing acceptance as a treatment option for chronic pain, there is little empirical research concerning long-term outcomes with this patient population. Several important questions concerning the use of opioids have yet to be examined in controlled studies. These include: determination of the most effective dosing regime, specification of the risk factors for medication abuse, and identification of patients most likely to achieve long-term benefits. Despite the lack of empirical data, the clinical literature to date yields two general approaches to the use of opioid treatment with chronic, nonmalignant pain. The first approach dictates that due to risk of addiction, tolerance, and insensitivity to large doses, opioid medications should be carefully controlled, with minimal and stable dosing as the eventual goal of treatment. The second approach, fostered by the beneficial use of opioids in the treatment of cancer pain, maintains that risk of addiction and abuse has been exaggerated. Proponents of this approach suggest that under-medication is a significant cause of treatment failure and non-compliance in chronic pain patients, and that prescription guidelines should emphasize patients� reports of adequate relief, regardless of dosage.

DETAILED DESCRIPTION:
BACKGROUND AND CLINICAL RELEVANCE: Although the use of opioid medications has gained increasing acceptance as a treatment option for chronic pain, there is little empirical research concerning long-term outcomes with this patient population. Several important questions concerning the use of opioids have yet to be examined in controlled studies. These include: determination of the most effective dosing regime, specification of the risk factors for medication abuse, and identification of patients most likely to achieve long-term benefits. Despite the lack of empirical data, the clinical literature to date yields two general approaches to the use of opioid treatment with chronic, nonmalignant pain. The first approach dictates that due to risk of addiction, tolerance, and insensitivity to large doses, opioid medications should be carefully controlled, with minimal and stable dosing as the eventual goal of treatment. The second approach, fostered by the beneficial use of opioids in the treatment of cancer pain, maintains that risk of addiction and abuse has been exaggerated. Proponents of this approach suggest that under-medication is a significant cause of treatment failure and non-compliance in chronic pain patients, and that prescription guidelines should emphasize patients' reports of adequate relief, regardless of dosage.

OBJECTIVES: The proposed study will test two core hypotheses:

1) What is the best overall approach to long-term (12 month) opioid therapy for chronic pain, and 2) Which of the potentially important predictor variables mentioned in the clinical opioid literature are related to outcome in an outpatient Veteran population.

RESEARCH PLAN AND METHODS: The two approaches to opioid use will be operationalized using medication prescription guidelines as two separate groups (Tolerable Pain Dosage vs. Adequate Relief Dosage) to be tested in a randomized trial. For the Tolerable Pain group, opioid medications will be prescribed at initially low doses with the expectation that low dosing will be adequate to reduce pain to a tolerable level. Dose increases are done slowly and only based on reports of some relief with low dose, with the goal of low and stable dosing to prevent dependence and tolerance. For the Adequate Relief group, opioid dosage is initially rapidly increased until the patient indicates adequate or substantial relief, at which point dosage is stabilized. For this group, tolerance and dependence are viewed as signs of inadequate dosing and handled typically with dose increases. Both groups will share some common guidelines such as monthly monitoring, random screens for other drug use, and prescriptions limited to a single clinic. Outcome will be measured with respect to primary outcome variables of pain relief, quality of life, and addictive behaviors, with secondary outcome variables of medication use, mood, illness beliefs, treatment satisfaction, and health care utilization. These variables will be assessed at study entry, and at 4 month, 8 month and 12 month follow-up visits. In addition, the following individual difference variables will be examined to determine patient characteristics that may impact on treatment outcome: psychosocial factors (e.g., history of substance abuse, economic status, environmental support), type and chronicity of pain problem, mood, medication use, quality of life, and illness impact. These variables will also be assessed at study entry and at 4 month, 8 month and 12 month follow-up visits.

PROGRESS REPORT AND CURRENT FINDINGS: Subject enrollment and follow-up has been completed, a total of 135 subjects were enrolled. Data analysis is ongoing. Primary hypotheses are being investigated in the current analyses and results are pending.

ELIGIBILITY:
Inclusion Criteria:

Veteran within Greater Los Angeles Healthcare System; Presence of chronic non-malignant pain for at least 6 months

Exclusion Criteria:

Anticipated surgery within 6 months; Current testing for pain etiology; Serious health conditions (pulmonary disease, congestive heart failure); Active or recent (past 2 years) substance abuse problems; Psychiatric hospitalization within past 2 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2001-08; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Measure: Pain Relief (Visual Analogue Scales of pain variables and relief measures); Measure: Quality of Life (Oswestry Disability Index); Measure: Addictive Behaviors (Prescription Drug Use Questionnaire, Addiction Behaviors Checklist, Reason for Opioid

SECONDARY OUTCOMES:
Medication Use; Stability of Use; Treatment Satisfaction; Mood; Illness Beliefs; Health Care Utilization

CONTACTS AND LOCATIONS:
Overall Officials: Bruce D Naliboff, PhD MA, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

REFERENCES:
- [Result] Divono EC, Singh M, Renner SW, Baria AM, Schieffer B, Korobkin S, Naliboff BD. Comparison of opiate test results obtained from the LX20, AxSYM, REMEDi HS and RapidOne Oxy testing systems with prescribed medications. Clinical Chemistry. 2003 May 1; 49(S6):A77.
- [Result] Naliboff BD, Wu SM, Pham Q. Clinical considerations in the treatment of chronic pain with opiates. J Clin Psychol. 2006 Nov;62(11):1397-408. doi: 10.1002/jclp.20319. PMID 16937352
- [Result] Wu SM, Compton P, Bolus R, Schieffer B, Pham Q, Baria A, Van Vort W, Davis F, Shekelle P, Naliboff BD. The addiction behaviors checklist: validation of a new clinician-based measure of inappropriate opioid use in chronic pain. J Pain Symptom Manage. 2006 Oct;32(4):342-51. doi: 10.1016/j.jpainsymman.2006.05.010. PMID 17000351